CLINICAL TRIAL: NCT02182050
Title: A Double-blind, Randomised Phase II Study to Determine Efficacy and Safety of Oral Treatment With BIBF 1120 ES 250 mg Twice Daily Versus 150 mg Twice Daily in Patients Suffering From Advanced Non-small-cell Lung Cancer
Brief Title: Efficacy and Safety of Oral Treatment With BIBF 1120 ES in Advanced Non-small-cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1199.10
Record Dates: First submitted 2014-07-02; First posted 2014-07-08 (Estimated); Last update posted 2017-12-28 (Actual); Status verified 2017-12

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

ARMS (3):
- BIBF 1120 ES low dose (Experimental)
  Interventions: Drug: BIBF 1120 ES low dose
- BIBF 1120 ES high dose (Experimental)
  Interventions: Drug: BIBF 1120 ES high dose
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo to BIBF 1120 ES

INTERVENTIONS:
Drug: BIBF 1120 ES low dose
  Arms: BIBF 1120 ES low dose
Drug: BIBF 1120 ES high dose
  Arms: BIBF 1120 ES high dose
Drug: Placebo to BIBF 1120 ES
  Arms: Placebo

SUMMARY:
The overall purpose of this phase II trial was to evaluate the efficacy of 250 mg BIBF 1120 twice daily (BID) versus 150 mg BIBF 1120 BID in patients with advanced non-small-cell lung cancer (NSCLC) who had failed at least one prior chemotherapy regimen. In addition, safety data for the two different dosages were collected and analysed.

ELIGIBILITY:
Inclusion criteria:

1. Male or female patients with histologically confirmed advanced NSCLC (i.e. adenocarcinoma, squamous cell carcinoma, large cell carcinoma, or combinations of these) stage IIIB (including pleural effusion) and stage IV.
2. Patients with recurrent disease who relapsed after previous treatment with platinum- or non-platinum based chemotherapy.
3. Full recovery from all therapy related toxicities from previous chemotherapy/ radiotherapy or recovery in as much as no further improvement may be expected by the investigator.
4. Age ≥18 years.
5. Life expectancy of at least 3 months.
6. ECOG performance score 0, 1 or 2.
7. Uni-dimensionally measurable tumour lesions by one or more techniques, i.e. CT, MRI, X-ray.
8. Adequate hepatic function: total bilirubin within normal limits; alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) ≤ 1.5x upper limit of normal (ULN) in patients without liver metastasis; For patients with liver metastasis: total bilirubin ≤ 1.5x ULN; ALT and/or AST < 2.5x ULN.
9. Coagulation parameters: international normalised ratio less than 1.3 or prothrombin time (PT) and partial thromboplastin time (PTT) less than 1.5 times institutional ULN.
10. Adequate renal function: serum creatinine ≤ 1.5 x upper normal limit.
11. Absolute neutrophil count (ANC) ≥ 1500/mL, platelets ≥ 100000/mL, haemoglobin ≥ 9.0 g/dL.
12. Written informed consent consistent with ICH-GCP guidelines and local law.

Exclusion criteria:

1. Active brain metastases stable for < 4 weeks, symptomatic, or requiring treatment with anti-convulsants and/or steroids or leptomeningeal disease.
2. Patients with history of haemorrhagic or thrombotic event (including transient ischemic attacks) in the past 12 months. Known inherited predisposition to thrombosis.
3. Concurrent therapeutic anticoagulation (except heparin flush as needed for maintenance of an indwelling intravenous device) or antiplatelet therapy (except chronic low-dose daily acetylsalicylic acid < 325mg).
4. Sanguineous pleural effusion due to disease or pericardial effusion suspicious for disease.
5. Clinically significant haemoptysis (1 teaspoon or more) within the last 3 months.
6. Centrally located tumours with radiographic evidence (CT or MRI) of local invasion of major blood vessels.
7. Radiographic evidence of cavitary or necrotic tumours at screening.
8. Major injuries and surgeries. Planned surgical procedures during the trial. Patients with incomplete wound healing within the past 4 weeks.
9. Gross haematuria within the last 3 months.
10. Significant cardiovascular diseases (i.e. uncontrolled hypertension, unstable angina, history of myocardial infarction within the past 6 months, serious cardiac arrhythmia, congestive heart failure according to New York Heart Association (NYHA) III or IV.
11. Serious illness or concomitant non-oncological disease such as neurologic-, psychiatric- or infectious disease or laboratory abnormality that may increase the risk associated with study participation or study drug administration and in the judgment of the investigator would make the patient inappropriate for entry into the study.
12. Gastrointestinal abnormalities that would interfere with intake or absorption of the study drug, prior surgical procedures affecting absorption, treatment for peptic ulcer disease within the last 6 months, active gastrointestinal bleeding unrelated to cancer (as evidenced by either hematemesis, hematochezia, or melena in the past 3 months and without endoscopic documented resolution), or malabsorption syndromes.
13. Other malignancy within the past 5 years (other than non-melanomatous skin cancer or cervical carcinoma in situ).
14. Treatment with other investigational drugs (elimination half life < 5 days) within the past 4 weeks before visit 2 or participation in another clinical trial within the past 4 weeks before start of therapy (visit 2) or concomitantly with this trial.
15. Treatment with chemo-, immuno-, hormonotherapy or with biologic response modifier within the past four weeks prior to treatment with the trial drug and during the trial.
16. Radiotherapy within the last 4 weeks prior start of treatment with the trial drug and radiotherapy to an area of measurable disease.
17. Hypersensitivity to BIBF 1120 ES or the excipients of the trial drug.
18. Male or female patients who are sexually active and unwilling to use a medically acceptable method of contraception prior to study entry and for the duration of study participation.
19. Pregnancy or breast feeding.
20. Known or suspected active alcohol or drug abuse.
21. Patients unable to comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2005-08; Primary Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Tumour response according to response evaluation criteria in solid tumours (RECIST) | baseline, every 6 weeks for an expected mean observation duration of 9 months
Time to tumour progression | baseline, every 6 weeks for an expected mean observation duration of 9 months

SECONDARY OUTCOMES:
Overall survival | mean observation duration of 9 months
European Organization for Research and Treatment (EORTC) Quality of Life Questionnaire (QLQ) (EORTC QLQ-C30) score | mean observation duration of 9 months
EORTC QLC lung cancer module (QLQ-LC13) score | mean observation duration of 9 months
Incidence and intensity of adverse events, graded by Common Terminology Criteria (CTCAE) 3.0 | mean observation duration of 9 months
Changes in safety laboratory parameters | mean observation duration of 9 months
Eastern Cooperative Oncology Group (ECOG) performance score | mean observation duration of 9 months
Changes in vital signs (body temperature, blood pressure, pulse rate, respiratory rate) | mean observation duration of 9 months
Maximum plasma concentration (Cmax) | pre-dose, 1, 2, and 3 hours after administration
Area under the curve (AUC) | pre-dose, 1, 2, and 3 hours after administration

REFERENCES:
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/21212157